CLINICAL TRIAL: NCT02005419
Title: A Phase II, Randomized, Double-blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of the Combination of Gemcitabine and Metformin in Treating Patients With Pancreatic Cancer After Curative Resection
Brief Title: Metformin Combined With Gemcitabine as Adjuvant Therapy for Pancreatic Cancer After Curative Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xian-Jun Yu (Other)
Responsible Party: Sponsor-Investigator, Xian-Jun Yu, M.D., Ph.D., Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MET1310128-2
Record Dates: First submitted 2013-11-24; First posted 2013-12-09 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Stage IA Pancreatic Adenocarcinoma; Stage IB Pancreatic Adenocarcinoma; Stage IIA Pancreatic Adenocarcinoma; Stage IIB Pancreatic Adenocarcinoma
Keywords: Pancreatic Cancer; Pancreatic Adenocarcinoma; Metformin; Gemcitabine; Adjuvant Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gemcitabine + placebo (Placebo Comparator): gemcitabine at 1000 mg/m^2 on days 1, 8, and 15; placebo at 2 g on days 1-28
  Interventions: Drug: Gemcitabine; Drug: placebo
- gemcitabine + metformin (Experimental): gemcitabine at 1000 mg/m^2 on days 1, 8, and 15; metformin at 2 g on days 1-28
  Interventions: Drug: Gemcitabine; Drug: Metformin

INTERVENTIONS:
Drug: Gemcitabine — Patients receive gemcitabine 1000 mg/m^2 (iv, 30 minutes) on days 1, 8, and 15 for 3 weeks, followed by one week without treatment, and also receive placebo (Arm I)/ metformin (Arm II) on days 1-28. Treatment repeats every 4 weeks for up to 6 circles in the absence of disease recurrence or unacceptable toxicity.
  Other Names: GEMZAR
Drug: Metformin — Metformin will be administered at a dose of 500 mg twice daily. If well tolerated, the dose will be increased to 1000 mg twice daily in the second week. Treatment repeats every 4 weeks (2 g on days 1-28) for up to 6 circles in the absence of disease recurrence or unacceptable toxicity.
  Other Names: glucophage
  Arms: gemcitabine + metformin
Drug: placebo — Placebo will be administered at a dose of 500 mg twice daily. If well tolerated, the dose will be increased to 1000 mg twice daily in the second week. Treatment repeats every 4 weeks (2 g on days 1-28) for up to 6 circles in the absence of disease recurrence or unacceptable toxicity.
  Arms: gemcitabine + placebo

SUMMARY:
Pancreatic cancer represents the most lethal of the common malignancies with a 5-year survival rate of less than 5%. For patients who are eligible for potentially curative resection, despite mortality and morbidity rates after surgery have improved, the recurrence rate is up to 85% within 2 years. Data from clinical trials indicate that adjuvant chemotherapy enhances 5-year survival to ~25% for patients who have undergone surgery to remove their tumor; and gemcitabine is the standard regimen of chemotherapy. Metformin is the first-line treatment for type 2 diabetes mellitus. Literatures reported that metformin might inhibit tumor growth by blocking some enzymes needed for cell growth. Some retrospective studies have revealed that diabetic patients taking metformin were less likely to develop pancreatic cancer. Additionally, pancreatic cancer patients treated with metformin showed a better survival than those without metformin. In this study, the researchers intend to investigate the activity and safety of the combination of gemcitabine and metformin in treating patients with pancreatic cancer that have removed by surgery.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment
* Age ≥ 18 years and ≤ 80 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have histologically confirmed pancreatic adenocarcinoma (or any mixed pathology if adenocarcinoma is predominant) after curative resection (R0). The pathological staging does not exceed the stage IIB.
* No tumor lesions are seen by abdominal and thoracic CT scan 4~8 weeks after surgery, and no serious adverse events are occurred during this period
* The expected survival after surgery ≥ 6 months
* White blood cell (WBC) ≥ 3 × 10^9/L; Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; Platelets (PLT) ≥ 100 × 10^9/L; Hemoglobin (Hgb) ≥ 9 g/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/ alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤ 2.5 × institutional upper limit of normal (ULN); Total bilirubin (TBIL) ≤ ULN; Creatinine (CRE) ≤ 1.5 × ULN
* Prothrombin time (PT) and international normalized ratio (INR) ≤ 1.5 × ULN
* Patients with diabetes (diagnosed after surgery) are eligible for this trial; all diabetic patients who are enrolled on this study should discuss the need to change their diabetes management regimen with their primary care physician or endocrinologist prior to enrollment
* Diabetic patients who are on metformin are eligible as long as they have been on metformin for less than 6 months (estimated 6 months or less duration of metformin therapy from start of metformin to enrollment on study)

Exclusion Criteria:

* Active second primary malignancy or history of second primary malignancy within the last 3 years
* Patients who have received any form of anti-tumor therapy before surgery, including chemotherapy, radiotherapy, interventional chemoembolization, radiofrequency ablation, and molecular targeted therapy
* Use of any other investigational agents
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, internal hemorrhage, pancreatic leakage, bile leakage, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of allergic reactions attributed to compounds of similar chemical or biological composition to metformin or gemcitabine
* Current use of metformin for more than 6 months prior to enrollment on study
* Metabolic acidosis, acute or chronic, including ketoacidosis
* Pregnant or nursing women
* Human immunodeficiency virus (HIV)-positive patients
* Patients who are unwilling or unable to comply with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival at one year after curative resection | From date of randomization (after curative resection) until the date of first documented recurrence or date of death from any cause, whichever came first, assessed 2 months during therapy and 3 months thereafter up to 24 months
  To evaluate the therapeutic efficacy of gemcitabine chemotherapy with versus without metformin hydrochloride in terms of recurrence-free survival in patients with pancreatic cancer at one year after curative resection. Computed tomography (CT) scan

SECONDARY OUTCOMES:
Overall survival after curative resection | From date of randomization (after curative resection) until the date of death from any cause, assessed one month during therapy and 3 months thereafter up to 24 months
  To evaluate the overall survival of patients (after curative resection) treated with this regimen. Outpatient visit, phone interview
Quality of life score after curative resection | One month during therapy and 3 months thereafter up to 24 months
  To evaluate the quality of life score of patients (after curative resection) treated with this regimen. Outpatient visit, phone interview
Number of grade 3 and 4 toxicities according to NCI CTCAE version 4.0 | One week during therapy and 3 months thereafter up to 24 months
  To evaluate the occurrence of grade 3 and 4 toxicities according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE; version 4.0) in patients treated with this regimen. The toxicity profile includes but not limits neutropenia, thrombocytopenia, peripheral neuropathy, hypoglycemia, metabolic acidosis (acute or chronic, including ketoacidosis), which will be summarized as the percentage of patients by type and grade according to treatment group. Outpatient visit, laboratory findings

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, M.D., Ph.D., Principal Investigator — Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Shanghai Pancreatic Cancer Institute; Pancreatic Cancer Institute, Fudan University. Shanghai, China.
Locations (1):
- Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, China